CLINICAL TRIAL: NCT06337253
Title: Seasonal Malaria Chemoprevention Rapid Assessment Study Mozambique
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MOZ202401
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Malaria,Falciparum; Chemoprevention
MeSH Terms: conditions — Malaria, Falciparum | interventions — Sulfadoxine; Pyrimethamine; Amodiaquine

STUDY DESIGN:
Intervention Model Description: The intervention in this study is the administration of one cycle of SPAQ medicines. SPAQ medicines procured by Malaria Consortium are from one of the 3 manufacturers with WHO prequalification, with whom Malaria Consortium has framework agreements: Tridem Pharma, S Kant Healthcare Ltd, or MacLeods Pharmaceuticals Ltd.
  Each monthly SMC cycle consists of one dispersible tablet of SP and three daily dispersible tablets of AQ. There are two doses of SPAQ: a lower dose for children aged three to <12 months, and a higher dose for children aged 12 to 59 months. For children aged 12 to 59 months, the dosage comprises a single dose of a full tablet of SP 500/25mg and three daily doses of a full tablet of AQ 153mg. Those aged three to <12 months are administered half the dose given to those aged 12 to 59 months, given as full dispersible tablets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention in this study is the administration of one cycle of SPAQ medicines. SPAQ medicines procured by Malaria Consortium are from Tridem Pharma, one of the three manufacturers with WHO prequalification, with whom Malaria Consortium has framework agreements.
  Each monthly SMC cycle consists of one dispersible tablet of SP and three daily dispersible tablets of AQ. There are two doses of SPAQ: a lower dose for children aged 3-12 months, and a higher dose for children aged 12 to 59 months. For children aged 12 to 59 months, the dosage comprises a single dose of a full tablet of SP 500/25mg and three daily doses of a full tablet of AQ 153mg. Those aged 3-12 months are administered half the dose given to those aged 12 to 59 months, given as full dispersible tablets.
  Interventions: Drug: Sulfadoxine/pyrimethamine plus amodiaquine

INTERVENTIONS:
Drug: Sulfadoxine/pyrimethamine plus amodiaquine — Seasonal Malaria Chemoprevention with SPAQ has not been trialed or introduced in Malawi yet. This intervention trial is different from others because of the location and because, traditionally, a full round of SMC with SPAQ that involves between 3-5 cycles is administered. Our trial is the first one that will only distribute one cycle of SMC with SPAQ. The data collected during the 42 days after SMC distribution will be used to estimate the medicines chemoprevention effectiveness at preventing malaria in children aged 3-59 months. This data, together with the resistance markers data will then be fed into a dynamical model that collaborators at Imperial College London have developed that will predic the potential impact of upscaling SMC in similar geographies.
  Other Names: SPAQ

SUMMARY:
Seasonal malaria chemoprevention (SMC) is a highly effective community-based intervention to prevent malaria infections caused by Plasmodium falciparum in areas where the burden of malaria is high and malaria transmission is seasonal. SMC is commonly seen as a success story in the Sahel region, however, there are regions in east and southern Africa where malaria transmission is seasonal, and the burden is high. However, the same decision-making frameworks that was used in the Sahel are unlikely to be applicable to east and southern Africa due to higher pre-existing resistance to the drugs used, seasonality heterogeneity, contextual difference, and unknown cost-effectiveness, amongst others. This study aims to estimate the chemoprevention efficacy, potential upscale impact, acceptability, and feasibility of SMC with sulfadoxine-pyrimenthamine + amodiaquine (SP+AQ) medicines in Niassa Province in Mozambique.

The study is divided into two separate components with different objectives which outputs feed into each other: a non-randomized controlled trial to estimate the chemoprevention efficacy of SP+AQ; and a qualitative study that will evaluate the feasibility and acceptability of the intervention.

These will be the first studies analysing the chemoprevention efficacy, feasibility, acceptability, and potential scale-up impact of SMC in Niassa Province, Mozambique The outcomes of these studies aim to guide future policy changes at local, national, and international levels and potentially allow for a historically successful program to expand in a sustained and cost-effective way beyond the Sahel region.

DETAILED DESCRIPTION:
Chemoprevention efficacy component

Outcomes. Primary outcomes of the CPES component are chemoprevention failure (a positive qPCR for P. falciparum parasites on day 28 after SP+AQ administration or P. falciparum positive slides at any time from day 7), prevalence of antimalarial resistance markers among chemoprevention failures and drug concentrations among chemoprevention failures. Secondary outcomes include uncomplicated malaria within the first 28 days since SP+AQ administration, participant's hospitalization within the first 28 days, severe malaria within the first 28 days , and severe anaemia levels comparisons at baseline and endline of our study period.

Sample size. Seasonal malaria chemoprevention must be well tolerated and highly effective to justify its deployment. It is therefore necessary to characterize failure (malaria breakthrough) rates accurately. A sample size of 500 children per study arm receiving SP+AQ will have 80% power to detect at least a 3% breakthrough infection rate by day 28 with a 95% confidence interval of ±1.5%, in settings where infection incidence is at least 6 infections or more per child per year and chemoprevention efficacy equals that in SMC trials in West Africa.

Recruitment and data collection. Participant selection will be carried on day 0 of the SMC implementation campaign by one trained inquirer and one phlebotomist (fieldworkers) that will follow the SMC community distributors. In each eligible household from both intervention and control arms one SMC eligible child will be selected to take part in the study . If the household has more than one SMC eligible child, only one will be randomly selected. The inquirer will be responsible for taking the informed consent form confirming the eligibility criteria that can be found below and assigning a unique ID number to each child. A baseline questionnaire will be administered to record sociodemographic data such as date of birth, gender, date of interview, and residence location. A thick blood smear will also be taken upon participant recruitment. Follow-up visits at timepoints 7, 14, 21, 28, 42 days post SMC-cycle start will be carried in selected households. The CHWs will invite the caregiver to bring their children to the health facility on the specific day to collect the blood samples. A short questionnaire exploring if the child received other treatment or experienced any disease since SP+AQ administration will be administered every time a sample is taken during the scheduled sample collection days (Day 0, 7, 14, 21, 28, 42). Heel (children aged 3-6 months) and finger (7-59 months) pricks will be collected for thick smears slides and DBS. Dose, weight, age, mid-upper arm circumference, tympanic temperature, location, time, and date will be recorded for each child on day 0, 7, 14, 21, 28 and day 42. All slides will be stained by using the Giemsa method within 24 hours of collection at the closest health facility and stored in a slide box with silica gel. Slides and DBS samples will be sent on to MORU in Bangkok, Thailand for sample analysis, where they will be analysed using qPCR methodology to detect drug concentrations, low-level sub microscopic parasitaemia and SP and AQ resistance markers.12 Drug concentration processing will take place for all SMC drugs on days 7, for sulfadoxine and AQ for day 28 and only for AQ for day 42 (as all the other drugs will have been metabolized by then ). Individual surveys on day 42 after the final DBS is taken will be conducted to determine if the child received other treatment or experienced illness over the past month of study implementation. In the event these children become febrile and receive a confirmed RDT between day 0 and day 42, they will have an additional DBS taken.

Data analysis. Once the samples have been analysed, the MORU laboratory will send the processed data back to the focal point at MC where the relevant mutations distributions and proportions will be analysed comparing parasitological efficacy between groups of mutations. Descriptive statistics of the intervention and control groups' drug levels will be calculated for the determination of any correlations with treatment outcomes, in particular drug concentrations on day 7. The focus will be on outliers with low levels of drug concentration based on the metrics described. Day 28 positivity will be correlated to antimalarial drug resistance genotype. Chemoprevention failure rates can be reported on as the cumulative failure rate using Kaplan-Meier analysis of the proportion. A time to event analysis will also be conducted to indicate duration of SMC infection protection afforded when looking at chemoprevention failures during follow up through slide and/or positive DBS samples.

Feasibility and acceptability component Outcomes. The outcomes of the qualitative study will be recorded experiences, opinions and perceptions surrounding SMC, that will be recorded and analysed through interviews and focus group discussions.

Sample size. The participants recruited for this study component will be purposefully selected and fall under four main groups: caregivers of children eligible for SMC (2 FGDs), community health workers involved in the administration of SMC (2 FGDs), community members of recognized importance and respect in areas where SMC is implemented such as community leaders (5 KIIs), and key informants involved in SMC implementation, programme management and policy making (4KIIs).The exact number of FGDs and KIIs will depend on data saturation in each of the implementation scenarios.

Recruitment and data collection. Key informants for IDIs will be purposefully identified during a stakeholder analysis done prior to the start of the study. For the FGDs, sensitisation meetings will be conducted in each village by the research coordinator and the county health official and head of villages to discuss the aims of the research, what it will involve and if they are willing to allow villagers to participate. Research assistants will visit villages and purposively recruit caregivers in consultation with village leaders based on availability and willingness to participate, as communicated to the village leader. CHWs will be purposively identified at HFs in collaboration with the head of the facility based on their availability and willingness to participate in an FGD. The FGDs will be conducted in a quiet and neutral space previously elected by the research team, and the research assistants will work with the community leaders to keep the space private for the duration of the FGD.

All interviews and FGDs will be audio recorded following participants' consent, and will then be transcribed and translated verbatim, or using equivalent translation where more appropriate for maintaining the integrity of meaning.

Data analysis. Data collection and analysis will be conducted iteratively, with data analysis beginning at the point of data generation. Participant recruitment and topic guides being adapted after piloting, to confirm or refute hypothesis based on emerging findings, and potential discrepancies from majority themes. Both inductive and deductive coding approaches will be used for thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Within 3 to 59 months
* Parents have provided written consent

Exclusion Criteria:

* Outside 3 to 59 months or age
* Parents have not provided written consent

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2024-05-26 (Estimated); Study Completion 2024-11-26 (Estimated)

PRIMARY OUTCOMES:
Chemoprevention failure | 42 days
  A positive qPCR for P. falciparum parasites on day 28 after SP+AQ administration or P. falciparum positive slides at any time from day 7

SECONDARY OUTCOMES:
Uncomplicated malaria within 28 days | 28 days
  A positive qPCR result for P. Falciparu, parasites within the first 28 days after SPAQ was administed

CONTACTS AND LOCATIONS:
Overall Officials: Sam Gudoi, Study Director — Malaria Consortium

IPD SHARING:
Plan to Share IPD: Undecided